CLINICAL TRIAL: NCT03961386
Title: Development of a Prototype FallsTalk Caregiver Resource System
Brief Title: FallsTalk Falls Prevention Program for Caregivers and Persons With Memory Loss or Dementia
Acronym: FT-C
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brookside Research & Development Company (Industry)
Collaborators: National Institute on Aging (NIA) (NIH); Alzheimer's Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FT-Cv1.1; R43AG058399 (NIH)
Record Dates: First submitted 2019-05-22; First posted 2019-05-23 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Falls (Accidents) in Old Age
Keywords: prevention

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FallsTalk-C (Experimental): FallsTalk CG intervention
  Interventions: Behavioral: FallsTalk-C; Behavioral: FallsTalk
- FallsTalk (Active Comparator): FallsTalk intervention
  Interventions: Behavioral: FallsTalk
- PostCardOnly (No Intervention): Postcard only- Control group

INTERVENTIONS:
Behavioral: FallsTalk-C — The FT-C experimental intervention involves two face-to-face visits including Initial and Follow-up Interviews, CG training, daily interaction with the PwD using a computer with FT-C software, weekly check-in calls, weekly postcard completion and monthly check-in calls for at least six months and up to one year.
  Arms: FallsTalk-C
Behavioral: FallsTalk — The FallsTalk intervention involves two face-to-face visits including Initial and Follow-up Interviews,CG training, daily interaction with the PwD, weekly check-in calls, weekly postcard completion and monthly check-in calls for at least six months and up to one year.
  Other Names: Attentional control- the same number of steps and an equivalent amount of time is devoted to these participants.
  Arms: FallsTalk; FallsTalk-C

SUMMARY:
This randomized-control trial involves dyads consisting of a family caregiver (CG) and a person with memory loss or dementia (PwD). The FallsTalk Caregiver Resource System (FT-C) intervention is administered by the CG, whose role is to modify their interactions with the PwD. FT-C will create a 3-way partnership between an Interventionist and the dyad, capitalizing on CG-PwD interactions. The PwD will be observed by the CG and both will be evaluated by the study team. Brief daily FT-C intervention by the CG will stimulate the PwD's awareness and individualized weekly CG- check-ins with the Interventionist will increase the CG's skills. Our hypothesis is that FT-C will increase PwD's awareness of personal fall threats and encourage new falls prevention behaviors, resulting in reduced fall rates.

DETAILED DESCRIPTION:
This is a single-site preliminary trial enrolling dyads in Western Washington state only.

ELIGIBILITY:
Caregiver (CG) Inclusion Criteria:

* residence in western Washington state
* minimum age= 18
* family CG
* primary CG
* some daily personal contact with Person with Dementia (PwD) for 1 month
* basic computer skills and telephone access
* able to commit to 6 month study.

Persons with Dementia (PwD) Inclusion Criteria:

* living at home with residence in western Washington state
* minimum age= 55
* at least one fall in last 6 months or regular loss of balance
* can ambulate at least 6 feet
* ability to communicate thoughts
* willingness to participate.

CG Exclusion Criteria:

* Professional CG (unless primary CG for family member)
* distance CG unable to be physically present with PwD daily for 1 month
* terminal illness with less than 6 months to live
* CG has significant memory loss.

PwD Exclusion Criteria:

* Residence outside of western Washington state
* Living in Residential care setting
* non-communicative
* terminal illness with less than 6 months to live
* wheel chair or bed bound.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-03-13 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Rate of falls | weekly for up to one year
  number of falls per month
Change of Residence | weekly for up to one year
  Report of change of primary residence

SECONDARY OUTCOMES:
Fall Threat Awareness | Pre-test- 5 clips at Initial interview; Post-test- 5 clips at Follow-up interview one month later
  Ability to identify potential fall risks in 10 standardized novel multimedia clips administered in random order
Activity-Specific Balance Confidence scale | Pre-test at Initial interview; Post-test at Follow-up interview one month later
  The Activity-Specific Balance Confidence scale is a standardized 16 item scale that measures an individual's self-efficacy about preventing a fall or loss of balance. The maximum score is 1600. Each item is scored from 0-100 with 0 indicating no confidence and 100 meaning complete confidence.
Caregiver Falls Prevention Concerns | Survey administered at study entry and Follow-up visit.
  Specific concerns identified by Caregiver with respect to preventing falls in the person they care for.
Burden Scale for Family Caregivers | BSFC is administered at Initial interview and Follow-up interview one month later.
  The Burden Scale for Family Caregivers is a standardized 28 item scale that assesses subjective burden of the CG. The items are scored as strongly agree, agree, disagree or strongly disagree and the maximum score is 84. A score of 0 indicates no burden and a score of 84 indicates a very severe burden with a high risk of psychosomatic symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Panzer, PhD, Principal Investigator — Brookside Research & Development
Locations (1):
- Brookside Research & Development, Freeland, Washington, United States

IPD SHARING:
Plan to Share IPD: No